CLINICAL TRIAL: NCT07290738
Title: TMS for Negative Symptoms in Schizophrenia Spectrum Disorders
Brief Title: Transcranial Magnetic Stimulation (TMS) for Negative Symptoms in Schizophrenia Spectrum Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-25-0694
Record Dates: First submitted 2025-11-26; First posted 2025-12-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- AG TMS (Experimental)
  Interventions: Device: TMS
- PFC sham (Sham Comparator)
  Interventions: Device: sham
- AG Sham (Sham Comparator)
  Interventions: Device: sham
- PFC TMS (Active Comparator)
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — A wire coil is held on the scalp. Brief electrical currents are passed through the coil and create one or more magnetic pulses that stimulate the brain. For each TMS session, bursts of 3 pulses at 50 Hz are repeated at 5 Hz as a train for 2seconds. The inter-train interval is 8 seconds. There are 20 trains lasting 192 seconds (600pulses) per session. The intensity of TMS stimulations is set to 80-120% of resting motor threshold(RMT).
  Arms: AG TMS; PFC TMS
Device: sham — Participants will receive total of 2 s of theta burst sham stimulation (TBS) trains repeated every 10 s for a total of 20 cycles (600 pulses). No actual magnetic stimulation will occur, still participant hears the TMS sound and a skin sensation
  Arms: AG Sham; PFC sham

SUMMARY:
The purpose of this study is to determine if repetitive transcranial magnetic stimulation (rTMS) applied to angular gyrus (AG) will improve negative symptoms and/or other psychosis symptoms in schizophrenia spectrum disorders (SSD) patients compared with prefrontal cortex (PFC) or sham.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent
* Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above 10.
* Is currently under the care of a licensed primary care provider or mental healthcare provider (e.g., psychiatrist, psychologist, nurse practitioner, licensed clinical social worker).
* Have negative symptoms as determined by BNSS score of 20 or more.
* Agrees to provide written permission, as requested, to allow any and all forms of communication between the investigators and study staff and any health care provider who currently provides and/or has provided service to the subject within two years of study enrollment

Exclusion Criteria:

* Persons with a first-degree relative with inherited epilepsy, seizure disorder, or seizures or persons who answer "yes" to any of the parts (A. - G.) of Question 3 of an epilepsy screening questionnaire.
* Taking > 400 mg clozapine/day and not on anti-seizure medication(s) with sufficient dose.
* Failed TMS screening questionnaire.
* Significant alcohol or other drug use (substance dependence within the recent months) or positive urine toxicology screen for substance not prescribed other than nicotine or marijuana dependence.
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, Central nervous System (CNS)infection or tumor, other significant brain neurological conditions.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* History of head injury with loss of consciousness over 10 minutes; history of brain surgery
* 0 Cannot refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
* Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive pregnancy test) or has had unprotected sexual intercourse without birth control in the last 4 weeks.
* Moderate-High Risk of suicide according to the Columbia - Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent (i.e. answers YES to Question 2 and NO to Question 6 (Moderate risk); or answers YES to Questions 3 (Moderate risk), 4, 5, or 6 (High risk) or in the clinical judgement of the investigator or the study psychiatrist.
* History (or family history) of deep vein thrombosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood-brain barrier (BBB) water exchange rate at AG obtained from MRI scan | baseline (before treatment visit 1), midpoint (after treatment visit 10; about 2 weeks from baseline), and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)

SECONDARY OUTCOMES:
Change in Negative symptoms as assessed by the Brief Negative Symptom Scale (BNSS) | at baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  It includes 13 items across 6 domains: blunted affect, alogia, asociality, anhedonia, avolition, and lack of normal distress. Each item is scored from 0 to 6, with higher scores indicating more severe negative symptoms.
  The total score ranges from 0 to 78.
Change in Positive symptoms as assessed by the Positive and Negative Syndrome Scale (PANSS) | at baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  It includes 30 items rated from 1 (absent) to 7 (extreme) across three subscales:
  Positive Symptoms (7 items; score range 7-49) Negative Symptoms (7 items; score range 7-49) General Psychopathology (16 items; score range 16-112) The PANSS Total Score ranges from 30 to 210, with higher scores indicating more severe symptoms. Change
Change in Cognitive function as assessed by Brief Assessment of Cognition in Schizophrenia (BACS): Symbol Coding | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Participants are asked to match symbols to numbers according to a key as quickly and accurately as possible within 90 seconds. Scores reflect the total number of correct responses, with higher scores indicating better cognitive performance.
Change in Working memory as assessed by the Number Span test | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  The Number Span test evaluates working memory capacity by requiring participants to recall sequences of numbers in the same order (forward span) and/or reverse order (backward span). Scores represent the total number of correctly recalled sequences, with higher scores indicating better working memory performance.
Change in Working memory as assessed by the Wechsler Memory Scale-Third Edition (WMS-III): Spatial Span | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Participants observe a series of blocks tapped by the examiner and are asked to reproduce the sequence in the same order (Spatial Span Forward) and reverse order (Spatial Span Backward).
  Scores are based on the number of correctly reproduced sequences, with higher scores indicating better spatial working memory performance.
Change in Cognitive function as assessed by the Category Fluency Test: Animal naming (Fluency) | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  participants are asked to name as many animals as possible within 60 seconds.
  The score is the total number of correct, non-repeated animal names, with higher scores indicating better semantic fluency.
Change in Cognitive function as assessed by the Rey-Osterrieth Complex Figure Test | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Participants are asked to copy a complex geometric figure and later reproduce it from memory after a delay.
  Scores are based on the accuracy and placement of figure components, with higher scores indicating better visuospatial and memory performance.
Change in Cognitive function as assessed by the Bell Lysaker Emotion Recognition Task | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Participants view brief video clips of an actor expressing various emotions (e.g., happiness, sadness, anger, fear, surprise, disgust, and neutrality) through facial expressions, vocal tone, and body language.
  Participants identify the emotion portrayed in each clip. Scores reflect the total number of correctly identified emotions, with higher scores indicating better emotion recognition ability.
Change in Cognitive function as assessed by the Hinting Task | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Participants read or listen to brief scenarios in which a character implies a desire or intention, and they must identify the underlying meaning.
  Scores reflect the total number of accurately interpreted hints, with higher scores indicating better theory of mind functioning.
Change in Depression as assessed by the Patient Health Questionnaire (PHQ-9) | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  The PHQ-9 is a 9-item self-report questionnaire that measures depressive symptom severity over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day), yielding a total score range of 0-27, with higher scores indicating more severe depression.
Change in Depression as assessed by the Calgary Depression Scale | t baseline, after treatment visit 10 (about 2 weeks from baseline), and at the end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Total score of the Calgary Depression Scale will be reported and ranges from 0 to 27, with a higher score indicating greater depression.
Change in Resting state functional connectivity between AG and PFC assessed by functional MRI (fMRI) | at baseline (before treatment visit 1), midpoint (after treatment visit 10; about 2 weeks from baseline), and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in Activity level (number of steps per day) as assessed by smart wristwatch | from baseline (before treatment visit 1) through end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in Location (number of unique places visited)as assessed by smart wristwatch | from baseline (before treatment visit 1) through end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in Sleep (number of hours slept per day) as assessed by smart wristwatch | from baseline (before treatment visit 1) through end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in Speech (pitch, intonation, pause) as assessed by video recording of speech | baseline, after treatment visit 10 (about 2 weeks from baseline), and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in facial expression (neutral, positive, and negative facial features) as assessed by video recording of speech | baseline, after treatment visit 10 (about 2 weeks from baseline), and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
Change in Electrophysiological responses as indicated by mismatch negativity as measured by electroencephalography (EEG) | baseline (before treatment visit 1) and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Mismatch negativity values will be reported in microvolts (uV). Mismatch negativity is measured by subtracting the averaged response to a set of standard stimuli from the average response to deviant stimuli, and taking the amplitude of this difference in a given timepoint.
Change in Electrophysiological response as indicated by steadystate auditory evoked responses from electroencephalography recording (EEG) | baseline (before treatment visit 1) and end of acute treatment (after treatment visit 20; about 4 weeks from baseline)
  Steady-state auditory evoked responses will be reported. The responses are measured by calculating the ratio of the power at target frequency over power at the surrounding background frequencies. The ration will be obtained in a given timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No